CLINICAL TRIAL: NCT05745922
Title: Acute Effects of Endurance Exercise With Moderate and High Intensity on Breast Milk Composition Among Women With Overweight/Obesity
Brief Title: Acute Effects of Endurance Exercise on Breast Milk Composition in Women With Overweight/Obesity
Acronym: YT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 562012
Record Dates: First submitted 2023-02-08; First posted 2023-02-27 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Breast Milk Collection; Overweight and Obesity
Keywords: Exercise
MeSH Terms: conditions — Breast Milk Expression; Overweight; Obesity; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Sequential assignment
Who Masked: Outcomes Assessor
Masking Description: The personnel who will be analysing the milk samples will be blinded to which condition the samples were obtained from and the time-point.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Resting in seated position
- Moderate intensity exercise (Experimental): Moderate intensity endurance exercise, treadmill walking/running at 70% of heart rate maximum for 40 minutes
  Interventions: Behavioral: Moderate intensity exercise
- High intensity exercise (Experimental): High intensity interval training: treadmill walking/running. 10 minutes warm-up at 70% of heart rate maximum, followed by four 4-minutes bouts at 90-95% of heart rate maximum, separated by 3-minutes active recovery (at 70% of heart rate maximum)
  Interventions: Behavioral: High intensity exercise

INTERVENTIONS:
Behavioral: Moderate intensity exercise — Treadmill walking/running with moderate intensity
  Arms: Moderate intensity exercise
Behavioral: High intensity exercise — Treadmill walking/running with high intensity
  Arms: High intensity exercise

SUMMARY:
The investigators will determine the acute effect of exercise on breastmilk composition. Participants will come in to the lab on three different days, out of which they will exercise on two of these days and rest in the lab on the third day. The conditions will be randomly allocated to each participant. Breastmilk samples will be obtained in the morning of each test day, as well as immediately after, one hour after and four hours after the exercise/rest condition. Dietary intake will be standardized on the test days.

ELIGIBILITY:
Inclusion Criteria:

* 6 weeks postpartum
* Exclusively breastfeeding
* Term birth
* Singleton baby

Exclusion Criteria:

* Known cardiovascular disease
* Known type 1 or type 2 diabetes
* Limited ability to exercise

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Breastmilk metabolite composition | Change from before exercise to after exercise (+0 hour, +1 hour, and +4 hours)
  Global metabolomics profiling using MS/MS technology

SECONDARY OUTCOMES:
Complex lipids composition | Change from before exercise to after exercise (+0 hour, +1 hour, and +4 hours)
  Global metabolomics profiling using MS/MS technology
Adiponectin | Change from before exercise to after exercise (+0 hour, +1 hour, and +4 hours)
  Concentration
Leptin | Change from before exercise to after exercise (+0 hour, +1 hour, and +4 hours)
  Concentration
Insulin Growth Factor-1 | Change from before exercise to after exercise (+0 hour, +1 hour, and +4 hours)
  Concentration
Insulin | Change from before exercise to after exercise (+0 hour, +1 hour, and +4 hours)
  Concentration
Ghrelin | Change from before exercise to after exercise (+0 hour, +1 hour, and +4 hours)
  Concentration
Cytokine profiling (Multiplex 27) | Change from before exercise to after exercise (+0 hour, +1 hour, and +4 hours)
  Concentration

OTHER OUTCOMES:
Cardiorespiratory fitness | At baseline
  Peak oxygen uptake
Body mass in kg | At baseline
  Impedance scale
Fat mass in kg | At baseline
  Impedance scale
Muscle mass in kg | At baseline
  Impedance scale
Height in metres | At baseline
  Stadiometer

CONTACTS AND LOCATIONS:
Locations (1):
- Department of circulation and medical imaging , NTNU, Trondheim, Norway

DOCUMENTS (4):
  • Study Protocol (2025-02-26): https://cdn.clinicaltrials.gov/large-docs/22/NCT05745922/Prot_000.pdf
  • Statistical Analysis Plan (2025-09-07): https://cdn.clinicaltrials.gov/large-docs/22/NCT05745922/SAP_001.pdf
  • Informed Consent Form: Partner (2024-01-02): https://cdn.clinicaltrials.gov/large-docs/22/NCT05745922/ICF_002.pdf
  • Informed Consent Form: Participant (mother) (2024-01-02): https://cdn.clinicaltrials.gov/large-docs/22/NCT05745922/ICF_003.pdf